CLINICAL TRIAL: NCT07159737
Title: Comparison of Hybrid Versus Two-Stent Strategies in Patients With Unprotected True Left Main Coronary Artery Bifurcation Disease: A Streamlined, Multicentre, Investigator-Initiated, Randomized Superiority Trial (HYBRID MAIN)
Brief Title: Comparison of HYBRID Versus Two-Stent Strategies in Unprotected True Left MAIN Bifurcation
Acronym: HYBRID MAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sultanah Bahiyah (Other Government)
Collaborators: Clinical Research Malaysia (Unknown)
Responsible Party: Principal Investigator, Dharmaraj Karthikesan, Consultant Interventional Cardiologist, Hospital Sultanah Bahiyah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81117075727
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Unprotected Left Main Coronary Artery Disease
Keywords: drug-eluting stent; drug-coated balloon; unprotected left main coronary artery disease; hybrid strategy; two-stent strategy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-stent strategy (Active Comparator): Detailed technique is described in the Detailed study description paragraph
  Interventions: Procedure: Two-stent strategy
- Hybrid strategy (Experimental): Detailed technique is described in the Detailed study description paragraph
  Interventions: Procedure: Hybrid Strategy

INTERVENTIONS:
Procedure: Two-stent strategy — DES from LMCA to LAD and DES to LCx using a recognised bifurcation technique such as double kissing crush (DK crush), Culotte, T-stenting or T and small protrusion (TAP).
  Arms: Two-stent strategy
Procedure: Hybrid Strategy — DES from LMCA to LAD and DCB to LCx. No LCx DES unless bail-out needed.
  Arms: Hybrid strategy

SUMMARY:
The number of deaths from heart disease is rising globally, particularly in developing countries. This condition involves the narrowing of arteries that supply blood to the heart. The most critical narrowing occurs in the left main coronary artery (LMCA), which supplies blood to over two-thirds of the heart muscle. Treating this narrowing is essential to prevent heart attacks or death. The LMCA divides into two branches, known as a bifurcation, both of which require treatment if narrowed.

Currently, narrowing in both branches-the left anterior descending artery (LAD) and the left circumflex artery (LCx)-is treated with a two-stent strategy, where metallic stents are placed in each branch to keep the arteries open. However, this approach is prone to re-narrowing, particularly at the origin of the LCx. A new procedure, called the hybrid strategy, offers an alternative. It involves placing one stent in the LMCA and LAD while inflating a special balloon in the LCX. This balloon, known as a drug-coated balloon, releases a chemical that reduces narrowing over time without needing a stent. At present, there is uncertainty which strategy is better. This study will assess whether the hybrid strategy is more effective than the two-stent strategy in preventing death, heart attacks, and re-narrowing of the arteries.

Participants will have an equal chance of receiving either the two-stent or hybrid strategy and will only join the study if their doctor is unsure which method is best. To minimise the burden on participants, all study procedures and follow-ups will be integrated into standard routine care.

The results of this study have the potential to offer a new, safer treatment that could save the lives of millions of people with this condition.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) of unprotected distal left main bifurcation (UTLMB) lesions remains technically demanding and is associated with higher risks than interventions in non-left main coronary lesions.

Several revascularisation strategies are in use:

* Provisional strategy - Implant a single drug-eluting stent (DES) from the left main coronary artery (LMCA) to the left anterior descending artery (LAD), leaving the left circumflex artery (LCx) unstented.
* Stepwise provisional strategy - Begin with the LMCA to LAD DES as in the provisional strategy, then implant a stent in the LCx only if required (e.g., for flow limitation or suboptimal angiographic result) using the operator's preferred method.
* Two-stent strategy - From the outset, plan to implant DES in both LAD and LCx using a recognised bifurcation technique.
* Hybrid strategy - Implant a DES from LMCA to LAD and treat the LCx with a drug-coated balloon (DCB) after adequate preparation and in the absence of a flow-limiting dissection.

While provisional approaches are less complex, they may be inadequate in true bifurcation lesions where both branches have significant disease.

Conversely, two-stent strategies offer full anatomical coverage but are technically challenging, associated with longer procedures, greater contrast use, higher radiation exposure, and potentially more periprocedural complications. Optimal outcomes heavily depend on the operator's skill, which contributes partly to the ongoing debate on this topic. Regardless of the operator's skill or chosen two-stent approach, the persistent risk of restenosis at the LCx ostium remains a significant vulnerability in the two-stent strategy.

The interventional cardiology community in the Asia-Pacific region remains divided on the optimal management of UTLMB due to differing philosophical and ideological approaches: the stepwise provisional strategy versus the upfront two-stent strategy. This uncertainty stems from conflicting results of two major RCTs focused on UTLMB.

The European Bifurcation Club MAIN (EBC MAIN) trial examined the stepwise provisional strategy, where a stent is placed from the LMCA to the LAD, and a second stent is added to the LCX only if necessary. Although underpowered, this trial found no significant difference in clinical outcomes at one year compared to the upfront two-stent strategy. However, recent three-year outcomes favour the stepwise provisional approach with lower repeat revascularisation rates.

Conversely, the DKCRUSH-V trial, conducted predominantly in Chinese centres with some sites outside China, compared an upfront two-stent strategy (double kissing crush [DK crush] technique) to a provisional strategy, showing better clinical outcomes at one year with the two-stent approach, with similar benefits at three years. The DK crush technique involves stenting the LCx first, followed by the LMCA to LAD.

The Hybrid Strategy, combining a DES and a DCB, has the potential to achieve full revascularisation while minimising metal implantation, preserving vessel compliance, and reducing late restenosis risk. Moreover, the hybrid strategy is technically less demanding and avoids the additional steps involved in the two-stent approach. Consequently, this approach is less dependent on the experience of the operator and can be more readily integrated into clinical practice. However, this approach has not yet been evaluated in a large-scale randomised controlled trial (RCT) for UTLMB lesions.

Asia-Pacific Perspective:

The burden of left main coronary artery disease is substantial in the Asia-Pacific region, where cardiovascular disease (CVD) remains the leading cause of mortality. Compared with Western populations, patients in this region often present with more diffuse and complex coronary artery disease (CAD). In many areas, there is limited availability of cardiothoracic surgeons, making PCI a more practical and timely option than coronary artery bypass graft surgery (CABG). There is also a strong patient preference for PCI over CABG, influenced by cultural factors, perceptions of surgical risk, and the shorter recovery time associated with PCI.

Interventional cardiology practice in the Asia-Pacific is characterised by high procedural volumes and substantial expertise in complex PCI techniques, including bifurcation stenting. DCBs are widely available and routinely used in parts of the region. These differences in patient characteristics, treatment preferences, procedural expertise, and technology access underpin the need for region-specific evidence.

The HYBRID MAIN trial has therefore been designed specifically for the Asia-Pacific setting, ensuring its findings will be directly relevant to the populations and healthcare systems most likely to benefit.

Primary Objective:

To determine whether a hybrid PCI strategy (DES from LMCA to LAD + DCB to LCx) is superior to an upfront two-stent strategy in reducing target lesion failure at 2 years in patients with UTLMB lesions suitable for both strategies

Trial Design:

The HYBRID MAIN trial is a streamlined, multicentre, open-label, randomised controlled trial (RCT) conducted exclusively in the Asia-Pacific region, testing the superiority of a hybrid strategy compared with an upfront two-stent strategy for UTLMB lesions.

Common principles:

* De novo UTLMB
* IVUS is mandatory for vessel sizing and lesion length before randomisation.
* LCx preparation must achieve residual stenosis < 30% without flow-limiting dissection.
* Operators preference to decide between upfront two-stent strategy or stepwise provisional approach

Eligible patients will be randomly allocated in a 1:1 ratio to receive either:

* Hybrid strategy: DES from the LMCA to the LAD with DCB to the LCx.
* Two-stent strategy: Implantation of DES in LMCA to the LAD and LCx using the operator's preferred bifurcation technique.

Pilot Phase:

The trial will commence with an internal pilot phase across selected high-volume PCI centres in Malaysia. The pilot will enrol the first 50 patients; if feasibility criteria are met, the trial will expand to multiple centres across the Asia-Pacific region.

Inclusion of High-volume Operators:

Only operators performing >300 PCI cases/year (including ≥20 left main interventions/year) will randomise patients. High-volume operators are more likely to apply the floating eligibility criteria effectively, achieve optimal procedural results, and minimise crossovers.

Recruitment:

Pre-screening performed by the operator based on diagnostic angiograms to determine whether the patient is potentially suitable for both strategies when substantial uncertainty exists. This aligns the trial with real-world decision-making and avoids unnecessary clinic visits for unsuitable cases.

Screening against the floating eligibility criteria, confirming:

* Unprotected distal LM true bifurcation (Medina 1,1,1; 1,0,1; and 0,1,1) with substantial uncertainty between both strategies
* Ability to give informed consent
* Pre-randomisation information

Written consent obtained before procedure wherever possible.

For patients identified during a coronary angiogram, urgent PCI may be required due to clinical indications or patient requests, with the operator deciding on the table. In these cases, pre-screening, screening, and consent occur simultaneously. For such cases, verbal consent may be obtained with written consent completed after the procedure.

After wiring both LAD and LCx;

* LAD and LCx vessel reference vessel diameter (RVD) and lesion length measured by IVUS before lesion preparation undertaken.
* Optimal lesion preparation in LCx with residual stenosis less than 30%, TIMI 3 flow without a flow-limiting dissection.
* May be part of stepwise provisional or upfront two-stent before randomisation.

Follow-up:

All patients will be followed for a mean of 2 years from the date of randomisation. Follow-up will be conducted by telephone or clinic visits, with medical record review as required. Post-trial follow-up will be done annually till 5 years post randomisation to look for long term clinical outcomes (TLF).

ELIGIBILITY:
Inclusion criteria:

Floating eligibility criteria

* De novo unprotected true left main bifurcation (UTLMB) (Medina 1,1,1; 1,0,1; and 0,1,1).
* Optimal LCx lesion preparation (residual stenosis less than 30% with absence of flow-limiting dissection).
* The operator feels it might be appropriate to place either a drug-eluting stent (DES) or drug-coated balloon (DCB) to the LCX
* Clinically stable at the time of randomisation.
* Able to complete 2-year follow-up.
* Able to complete dual antiplatelet therapy (DAPT) as per guidelines.
* Written informed consent (or verbal consent on-table with written consent as soon as possible thereafter).

Exclusion Criteria:

* Protected left main (patent graft to LAD and LCX)
* Need for anticoagulation
* LCx reference vessel diameter less than 2.5 mm (< 2.5 mm)
* Cardiogenic shock
* Severe left ventricular (LV) dysfunction making either strategy unsafe
* Contraindication to antiplatelet therapy or study devices
* Life expectancy less than 2 years
* Participation in another trial that may affect results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 2 years
  Target lesion failure (TLF) at 2 years defined as a composite of: time to first event of cardiovascular death, time to first event of target vessel myocardial infarction (TVMI), time to first event of clinically driven target lesion revascularisation (CD-TLR).

SECONDARY OUTCOMES:
Individual components of primary endpoint | 2 years
  Time to first event of individual components of TLF
  * time to first event of cardiovascular death
  * time to first event of TVMI
  * time to first event of CD-TLR
Composite of cardiovascular death and TVMI | 2 years
  Composite of objective endpoints included in TLF
  * time to first event of cardiovascular death
  * time to first event of TVMI
Safety endpoints | 2 years
  Time to first event of stent/lesion thrombosis

OTHER OUTCOMES:
Total procedure time | Immediately after the procedure
  Total procedure time defined as arterial puncture to completion of PCI
Contrast volume | Immediately after the procedure
  Total contrast volume used (mL)
Fluoroscopy dose | Immediately after the procedure
  Total fluroscopy dose using standard definition

CONTACTS AND LOCATIONS:
Overall Officials: Dharmaraj Karthikesan, M.D, MSc (Oxon), Principal Investigator — Hospital Sultanah Bahiyah, Alor Setar, Malaysia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Vervoort D, Lee G, Lin Y, Contreras Reyes JR, Kanyepi K, Tapaua N. 6 Billion People Have No Access to Safe, Timely, and Affordable Cardiac Surgical Care. JACC Adv. 2022 Aug 26;1(3):100061. doi: 10.1016/j.jacadv.2022.100061. eCollection 2022 Aug. No abstract available. PMID 38938403
- [Background] Rathore S, Tehrani S, Prvulovic D, Araya M, Lefevre T, Banning AP, Burzotta F, Rigatelli G, Gutierrez-Chico JL, Bonaventura K, Chevalier B, Kinoshita Y, Sikic J, Alfonso F, Louvard Y, Stankovic G. Drug coated balloons and their role in bifurcation coronary angioplasty: appraisal of the current evidence and future directions. Expert Rev Med Devices. 2020 Oct;17(10):1021-1033. doi: 10.1080/17434440.2020.1831385. Epub 2020 Oct 14. PMID 33000952
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Chen X, Li X, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Santoso T, Paiboon C, Kwan TW, Sheiban I, Leon MB, Stone GW, Chen SL; DKCRUSH-V Investigators. 3-Year Outcomes of the DKCRUSH-V Trial Comparing DK Crush With Provisional Stenting for Left Main Bifurcation Lesions. JACC Cardiovasc Interv. 2019 Oct 14;12(19):1927-1937. doi: 10.1016/j.jcin.2019.04.056. Epub 2019 Sep 11. PMID 31521645
- [Background] Loh PH, Lassen JF, Jepson N, Koo BK, Chen S, Harding SA, Hu F, Lo S, Ahmad WAW, Ye F, Guagliumi G, Hiremath MS, Uemura S, Wang L, Whelan A, Low A. Asia Pacific consensus document on coronary bifurcation interventions. EuroIntervention. 2020 Oct 9;16(9):e706-e714. doi: 10.4244/EIJ-D-19-00977. PMID 32250248
- [Background] Zhang JJ, Ye F, Xu K, Kan J, Tao L, Santoso T, Munawar M, Tresukosol D, Li L, Sheiban I, Li F, Tian NL, Rodriguez AE, Paiboon C, Lavarra F, Lu S, Vichairuangthum K, Zeng H, Chen L, Zhang R, Ding S, Gao F, Jin Z, Hong L, Ma L, Wen S, Wu X, Yang S, Yin WH, Zhang J, Wang Y, Zheng Y, Zhou L, Zhou L, Zhu Y, Xu T, Wang X, Qu H, Tian Y, Lin S, Liu L, Lu Q, Li Q, Li B, Jiang Q, Han L, Gan G, Yu M, Pan D, Shang Z, Zhao Y, Liu Z, Yuan Y, Chen C, Stone GW, Han Y, Chen SL. Multicentre, randomized comparison of two-stent and provisional stenting techniques in patients with complex coronary bifurcation lesions: the DEFINITION II trial. Eur Heart J. 2020 Jul 14;41(27):2523-2536. doi: 10.1093/eurheartj/ehaa543. PMID 32588060
- [Background] Chen SL, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Jiang T, Tao L, Zeng H, Li L, Xia Y, Gao C, Santoso T, Paiboon C, Wang Y, Kwan TW, Ye F, Tian N, Liu Z, Lin S, Lu C, Wen S, Hong L, Zhang Q, Sheiban I, Xu Y, Wang L, Rab TS, Li Z, Cheng G, Cui L, Leon MB, Stone GW. Double Kissing Crush Versus Provisional Stenting for Left Main Distal Bifurcation Lesions: DKCRUSH-V Randomized Trial. J Am Coll Cardiol. 2017 Nov 28;70(21):2605-2617. doi: 10.1016/j.jacc.2017.09.1066. Epub 2017 Oct 30. PMID 29096915
- [Background] Hildick-Smith D, Egred M, Banning A, Brunel P, Ferenc M, Hovasse T, Wlodarczak A, Pan M, Schmitz T, Silvestri M, Erglis A, Kretov E, Lassen JF, Chieffo A, Lefevre T, Burzotta F, Cockburn J, Darremont O, Stankovic G, Morice MC, Louvard Y. The European bifurcation club Left Main Coronary Stent study: a randomized comparison of stepwise provisional vs. systematic dual stenting strategies (EBC MAIN). Eur Heart J. 2021 Oct 1;42(37):3829-3839. doi: 10.1093/eurheartj/ehab283. PMID 34002215
- [Background] Dabrowski EJ, Kozuch M, Dobrzycki S. Left Main Coronary Artery Disease-Current Management and Future Perspectives. J Clin Med. 2022 Sep 28;11(19):5745. doi: 10.3390/jcm11195745. PMID 36233613